CLINICAL TRIAL: NCT03753958
Title: Antimicrobial Photodynamic Therapy Mediated by Papain Gel on Peri-implantitis Lesions: A Randomized Controlled Clinical Trial
Brief Title: Antimicrobial Photodynamic Therapy Mediated by Papain Gel on Peri-Implantitis Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Renato Araujo Prates, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bia
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe for measurements of plaque index, probing bleeding, probing depth, gingival recession and loss of clinical insertion. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT. The evaluator will not know to which group the patient belongs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): The treatment will consist of oral hygiene orientation, with brushing technique instructions and daily flossing recommendation. All patients will receive a demonstration of oral hygiene techniques. The calculus deposits on the teeth will be removed with an ultrasound equipment and curettes for root scaling and straightening13. In implants, calculus will be removed with specific curettes for use on the implant surface. Treatment will be performed in 2 to 4 sessions under local anesthesia (typically 2% mepivacaine with 1: 100,000 noradrenaline). Gracey periodontal curettes (numbers 3/4, 7/8, 11/12 and 13/14) and Mc Call for removal of the dental calculus will be used. Other biofilm-retaining factors, such as carious lesions, condemned teeth and maladaptive restorations, will be removed during these periodontal treatment sessions.
  Interventions: Procedure: Conventional treatment
- aPDT group (Experimental): aPDT will be performed after conventional treatment, in sites with pockets greater than or equal to 5 mm. The PapaMblue® photosensitizer with 100 μM methylene blue will be deposited in the pockets with a syringe, with the bottom of the pouch in the coronal direction, and a pre-irradiation time of 1 min will be adopted, so that the PS may stain the entire bacterial biofilm. Then, the laser emitting an wavelength of 660 nm, with power of 100 mW, will be applied. The laser will be applied to the mucosa on the oral epithelium with an optical fiber (apparatus of DMC Therapy EC, São Carlos, Brazil). Irradiation will be performed until the entire peri-implanted pouch is illuminated for 2 minutes at each point. The 6 points around the implant will be irradiated and each irradiation point will present an area of 0.4 cm2, which will result in radiant exposure of 30 J/cm2 following 2 min of irradiation per point. The irradiation will have a constant power density of 250 mW/cm2.
  Interventions: Procedure: Conventional treatment; Radiation: aPDT

INTERVENTIONS:
Procedure: Conventional treatment — The treatment will consist of oral hygiene orientation, with brushing technique instructions and daily flossing recommendation. All patients will receive a demonstration of oral hygiene techniques. The calculus deposits on the teeth will be removed with an ultrasound equipment and curettes for root scaling and straightening13. In implants, calculus will be removed with specific curettes for use on the implant surface. Treatment will be performed in 2 to 4 sessions under local anesthesia. Other biofilm-retaining factors, such as carious lesions, condemned teeth and maladaptive restorations, will be removed during these periodontal treatment sessions.
Radiation: aPDT — aPDT will be performed after conventional treatment, in sites with pockets greater than or equal to 5 mm. The PapaMblue® photosensitizer with 100 μM methylene blue will be deposited in the pockets with a syringe, with the bottom of the pouch in the coronal direction, and a pre-irradiation time of 1 min will be adopted, so that the PS may stain the entire bacterial biofilm. Then, the laser emitting an wavelength of 660 nm, with power of 100 mW, will be applied. The laser will be applied to the mucosa on the oral epithelium with an optical fiber (apparatus of DMC Therapy EC, São Carlos, Brazil). Irradiation will be performed until the entire peri-implanted pouch is illuminated for 2 minutes at each point. The 6 points around the implant will be irradiated and each irradiation point will present an area of 0.4 cm2, which will result in radiant exposure of 30 J/cm2 following 2 min of irradiation per point. The irradiation will have a constant power density of 250 mW/cm2.
  Arms: aPDT group

SUMMARY:
The elimination of pathogenic microorganisms from the muco-gingival tissue and implant pockets system is one of the main aspects for success in the treatment of peri-implantitis. The purpose of this study is to conduct a blinded and randomized clinical trial to evaluate the effectiveness of photodynamic therapy in the treatment of peri-implantitis. Twenty implants with peri-implantitis will be selected. Implants will be randomly divided into two groups (n = 10), Group 1: control - conventional treatment and Group 2: conventional treatment and antimicrobial photodynamic therapy (aPDT). aPDT will be performed after the purse removal service in sites with pockets greater than or equal to 5 mm. The photosensitizer will be PapaMblue®, which will be deposited in the peri-implant pockets, with pre-irradiation time of 1 min. Next, the laser emitting a wavelength of 660 nm, with power of 100 mW, for 2 min, radiant exposure of 30 J/cm2 and power density of 250 mW/cm2 in the buccal and mesial regions will be applied. The distribution of the data within each group will be evaluated and the variances will be checked to choose a more appropriate statistical analysis. The sample calculation is based on the literature and the significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Have peri-implantitis;
* Have at least one implant with a clinical depth of probing equal to or greater than 5 mm;
* Age range of 18 to 65 years.

Exclusion Criteria:

* Smokers or ex-smokers who stopped the habit less than 12 months before the screening;
* Have decompensated diabetes;
* Anemia;
* Cancer;
* Pregnant;
* Use antibiotics in the last 3 months12;
* Make use of anti-inflammatories or have coagulation disorders (use of anticoagulants, presence of liver diseases, thrombocytopenia, immunosuppression);
* In orthodontic treatment;
* Patients who maintained a biofilm index higher than 25%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2019-12-02 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in plaque index | Baseline, 30 days and 60 days after treatment.
  For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of plaque index. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT.
Change in probing bleeding | Baseline, 30 days and 60 days after treatment.
  For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of probing bleeding. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT.
Change in probing depth | Baseline, 30 days and 60 days after treatment.
  For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of probing depth. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT.
Change in gingival recession | Baseline, 30 days and 60 days after treatment.
  For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of gingival recession. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT.
Change in loss of clinical insertion | Baseline, 30 days and 60 days after treatment.
  For the evaluation of clinical parameters, a single trained, calibrated examiner will examine 6 sites of each implant with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of loss of clinical insertion. The evaluation will be performed at the beginning of treatment, 30 and 60 days after the first application of aPDT.

SECONDARY OUTCOMES:
Microbiological examination (change in CFUs (Colony Forming Units)) | Baseline and immediately after treatment.
  The microbiological examination will be performed from subgingival biofilm samples collected from the mesial region of the peri-implant pockets of the selected implants. Two collections will be performed at each experimental site before and immediately after the aPDT and irradiation procedures. For the collection of the subgingival biofilm, a relative isolation of the teeth with cotton rollers will be performed, the supra-gingival biofilm will be removed with sterile gauze, and the subgingival biofilm sample will be obtained by inserting a sterile absorbent paper tip (no. 30) into the inside of the peri-implant pocket, being held in place for 30 s. The tips will be removed and stored in properly identified sterile plastic microtubes, with each paper cone being stored in a different microtube.
  The samples will be used to determine the CFUs (Colony Forming Units).